CLINICAL TRIAL: NCT02207907
Title: A Six Month Clinical Study Based in the US to Evaluate the Efficacy and Tolerability of Sodium Bicarbonate Toothpaste
Brief Title: To Evaluate the Efficacy and Tolerability of Sodium Bicarbonate Toothpaste
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202192; RH02433 (Other: GSK)
Record Dates: First submitted 2014-07-31; First posted 2014-08-04 (Estimated); Results first posted 2017-02-17 (Actual); Last update posted 2017-04-13 (Actual); Status verified 2016-12

CONDITIONS: Oral Hygiene
MeSH Terms: interventions — Sodium Bicarbonate; Sodium Fluoride

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sodium bicarbonate plus sodium fluoride (Experimental): Experimental dentifrice containing sodium bicarbonate plus 1150 parts per million (ppm) fluoride as sodium fluoride
  Interventions: Drug: Sodium bicarbonate plus sodium fluoride
- Sodium fluoride (Active Comparator): Toothpaste containing 1100 ppm fluoride as sodium fluoride
  Interventions: Drug: Sodium fluoride

INTERVENTIONS:
Drug: Sodium bicarbonate plus sodium fluoride — Experimental dentifrice containing sodium bicarbonate plus 1150 parts per million (ppm) fluoride as sodium fluoride
  Arms: Sodium bicarbonate plus sodium fluoride
Drug: Sodium fluoride — Toothpaste containing 1100 ppm fluoride as sodium fluoride
  Arms: Sodium fluoride

SUMMARY:
The primary objectives of this study will be to compare the Gingival Bleeding and Gingival Inflammation following twice daily use of a sodium bicarbonate experimental dentifrice compared to a 0% sodium bicarbonate toothpaste after 24 weeks of use. The study will be conducted at Silverstone Research Group. Participants will be recruited from their database and by use of an external recruitment agency.

ELIGIBILITY:
Inclusion Criteria:

* Good general health with (in the opinion of the investigator) no clinically significant and relevant abnormalities of medical history or oral/dental examination.
* A minimum of 20 permanent gradable teeth
* Moderate gingivitis present at the screening visit in the opinion of the investigator
* A total of 20 bleeding sites or greater at baseline visit
* Positive response to bleeding on brushing present at the screening visit

Exclusion Criteria:

* Pregnant or breast feeding women
* Tobacco chewers
* Current or relevant history of any serious, severe or unstable physical or psychiatric illness or any other medical condition (e.g. Diabetes Mellitus) that would make the participant unlikely to fully complete the study or any that increases the risk to the participants or undermines the data validity.
* Recent history (within the last year) of alcohol or other substance abuse
* Participants requiring prophylactic antibiotic treatment prior to dental therapy
* Known or suspected intolerance or hypersensitivity to the study materials (or closely related compounds) or any of their stated ingredients
* Have current active caries or any medical conditions which may directly influence gingival bleeding
* Use of concomitant or any systemic medication that, in the opinion of the investigator, might interfere with the outcome of the study or have an effect on gingival conditions within 14 days of gingival examinations
* Excessive calculus present that interferes with the probing examination for Gingival Bleeding Index
* Participation in another clinical study or receipt of an investigational drug or oral care product within 30 days of the screening visit
* An employee of the sponsor or the study site or members or their immediate family.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 247 (Actual)
Dates: Start 2014-08; Primary Completion 2015-02 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Las Vegas, Nevada, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The participants were recruited at a clinical site in the USA.
Groups:
- Sodium Bicarbonate Dentrifice: Experimental dentifrice containing sodium bicarbonate plus 1150 parts per million (ppm) fluoride as sodium fluoride
- 0% Sodium Bicarbonate Dentrifice: Toothpaste containing 1100 ppm fluoride as sodium fluoride
Period: Overall Study
Arm/Group | Sodium Bicarbonate Dentrifice | 0% Sodium Bicarbonate Dentrifice
Started | 124 | 123
Completed | 113 | 115
Not Completed | 11 | 8
Not completed — Lost to Follow-up | 3 | 1
Not completed — Withdrawal by Subject | 5 | 6
Not completed — Did not meet study criteria | 3 | 0
Not completed — Pregnancy | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sodium Bicarbonate Dentrifice | 0% Sodium Bicarbonate Dentrifice | Total
Number analyzed (Participants) | 124 | 123 | 247
Age, Continuous [Mean (Standard Deviation); unit: Years] | 34.52 (13.162) | 37.55 (13.977) | 36.03 (13.631)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69 | 72 | 141
  Male | 55 | 51 | 106

OUTCOME MEASURES:

1. Primary Outcome: Number of Gingival Bleeding Sites at 24 Weeks
Description: Number of gingival bleeding sites were measured as bleeding index via a single examiner using a color coded periodontal probe. The probe was engaged approximately 1 millimetre (mm) into the gingival crevice. A moderate pressure was used whilst sweeping from interproximal to interproximal along the sulcular epithelium. The BI scoring system used to measure bleeding sites is as follows: 0= No bleeding after 30 seconds; 1= Bleeding upon probing after 30 seconds; 2= Immediate bleeding observed. A bleeding site was considered as a BI score of 1 or 2.
Time Frame: Baseline, 24 weeks
Population: Intent-to-Treat (ITT) population, defined as those participants who received study treatment and had at least one post-baseline efficacy measurement.
Measure: Mean (Standard Error); unit: number of gingival bleeding sites
Arm/Group | Sodium Bicarbonate Dentrifice | 0% Sodium Bicarbonate Dentrifice
Number analyzed (Participants) | 118 | 122
number of gingival bleeding sites
  Number of Bleeding Sites at Baseline | 45.13 (1.393) | 45.84 (1.448)
  Number of Bleeding sites after 24 weeks | 18.67 (1.142) | 36.39 (1.510)
Statistical Analysis 1: Comparison: Sodium Bicarbonate Dentrifice vs 0% Sodium Bicarbonate Dentrifice; Test type: Superiority or Other; p < 0.0001, ANCOVA; From ANCOVA analysis with treatment group and smoking status as factors and baseline MGI and BI as covariates; Adjusted Mean Difference = -17.491, 95% CI 2-sided [-20.317 to -14.664] — Difference is first named treatment minus second named treatment such that a negative difference favors the first named treatment

2. Primary Outcome: Modified Gingival Index (MGI) at 24 Weeks
Description: The Modified Gingival Index (MGI) was assessed on facial and lingual surfaces at two sites on each tooth (papillae and margin). The scoring of the MGI was performed under dental office conditions using a standard dental light for illuminating the oral cavity. Compressed air, water and mouth mirrors were available to each examiner. This procedure was performed by a single examiner. The MGI scoring system is as follows: 0 = absence of inflammation; 1 = mild inflammation; slight change in color, little change in color; little change in texture of any portion of the marginal or papillary gingival unit; 2 = mild inflammation; criteria as above but involving the entire marginal or papillar gingival units; 3= moderate inflammation; glazing, redness, edema, and/ or hypertrophy of the marginal or papillary gingival unit; 4 = severe inflammation; marked redness, edema and/or hypertrophy of the marginal or papillary gingival unit, spontaneous bleeding, congestion, or ulceration
Time Frame: Baseline, 24 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Sodium Bicarbonate Dentrifice | 0% Sodium Bicarbonate Dentrifice
Number analyzed (Participants) | 118 | 122
Units on a scale
  Modified Gingival Index at Baseline | 2.53 (0.017) | 2.54 (0.018)
  Modified Gingival Index after 24 weeks | 2.23 (0.021) | 2.43 (0.210)
Statistical Analysis 1: Comparison: Sodium Bicarbonate Dentrifice vs 0% Sodium Bicarbonate Dentrifice; Test type: Superiority or Other; p < 0.0001, ANCOVA; From ANCOVA analysis with treatment group and smoking status as factors and baseline MGI and BI as covariates; Adjusted Mean Difference = -0.201, 95% CI 2-sided [-0.237 to -0.165] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Number of Gingival Bleeding Sites at 6 and 12 Weeks.
Description: as for outcome 1
Time Frame: Baseline, 6 and 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: number of gingival bleeding sites
Groups:
- 0% Sodium Bicarbonate: Toothpaste containing 1100 ppm fluoride as sodium fluoride
Arm/Group | Sodium Bicarbonate Dentrifice | 0% Sodium Bicarbonate
Number analyzed (Participants) | 118 | 122
number of gingival bleeding sites
  Number of Bleeding Sites at Baseline | 45.13 (1.393) | 45.84 (1.448)
  Number of Bleeding Sites after 6 weeks | 25.40 (0.999) | 40.27 (1.448)
  Number of Bleeding sites after 12 weeks | 20.83 (0.915) | 34.23 (1.260)

4. Secondary Outcome: Modified Gingival Index (MGI) at 6 and 12 Weeks.
Description: MGI was assessed on facial and lingual surfaces at two sites on each tooth (papillae and margin). The scoring of the MGI was performed under dental office conditions using a standard dental light for illuminating the oral cavity. Compressed air, water and mouth mirrors were available to each examiner. This procedure was performed by a single examiner. The MGI scoring system is as follows: 0 = absence of inflammation; 1 = mild inflammation; slight change in color, little change in color; little change in texture of any portion of the marginal or papillary gingival unit; 2 = mild inflammation; criteria as above but involving the entire marginal or papillar gingival units; 3= moderate inflammation; glazing, redness, edema, and/ or hypertrophy of the marginal or papillary gingival unit; 4 = severe inflammation; marked redness, edema and/or hypertrophy of the marginal or papillary gingival unit, spontaneous bleeding, congestion, or ulceration
Time Frame: Baseline, 6 and 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Sodium Bicarbonate Dentrifice | 0% Sodium Bicarbonate Dentrifice
Number analyzed (Participants) | 118 | 122
Units on a scale
  Modified Gingival Index at Baseline | 2.53 (0.017) | 2.54 (0.018)
  Modified Gingival Index after 6 weeks | 2.28 (0.017) | 2.45 (0.018)
  Modified Gingival Index after 12 weeks | 2.24 (0.018) | 2.40 (0.018)

5. Secondary Outcome: Bleeding Index at 6, 12 and 24 Weeks
Description: The Bleeding Index was performed by a single examiner using a color coded periodontal probe. The probe was engaged approximately 1 millimetre (mm) into the gingival crevice. A moderate pressure was used whilst sweeping from interproximal to interproximal along the sulcular epithelium. The BI scoring system to be used is as follows: 0= No bleeding after 30 seconds; 1= Bleeding upon probing after 30 seconds; 2= Immediate bleeding observed
Time Frame: Baseline, 6, 12 and 24 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Units on a Scale
Arm/Group | Sodium Bicarbonate Dentrifice | 0% Sodium Bicarbonate Dentrifice
Number analyzed (Participants) | 118 | 122
Units on a Scale
  Bleeding Index Score at Baseline | 0.45 (0.014) | 0.47 (0.014)
  Bleeding Index Score after 6 weeks | 0.25 (0.010) | 0.41 (0.014)
  Bleeding Index Score after 12 weeks | 0.21 (0.009) | 0.35 (0.012)
  Bleeding Index Score after 24 weeks | 0.19 (0.012) | 0.37 (0.014)

6. Secondary Outcome: Plaque Control (Overall and Interproximal Dental Plaque Scores) Using Turesky Modification of Quigley &Amp; Hein Plaque Index at 6, 12 and 24 Weeks.
Description: The dental examiner used the Turesky Modification of the Quigley Hein Index to assess plaque on all gradable teeth. The plaque was first disclosed using a dye solution. Participants then rinsed with disclosing solution according to instructions. They had expectorated and rinsed with 10 mL of water for 10 seconds and expectorated again. Plaque was assessed with each tooth being divided into 6 areas including the mesiofacial, facial, distofacial, mesiolingual, lingual and distolingual surfaces. Disclosed plaque was scored as follows: 0= No plaque; 1= Slight flecks of plaque at the cervical margin of the tooth; 2= A thin continuous band of plaque (1 mm or smaller) at the cervical margin of the tooth; 3= A band of plaque wider than 1 mm but covering less than 1/3 of the crown of the tooth; 4= Plaque covering at least 1/3 but less tan 2/3 of the crown of the tooth; 5= Plaque covering 2/3 or more of the crown of the tooth
Time Frame: Baseline, 6,12 and 24 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Sodium Bicarbonate Dentrifice | 0% Sodium Bicarbonate Dentrifice
Number analyzed (Participants) | 118 | 122
Units on a scale
  Overall Plaque Score at Baseline | 3.04 (0.019) | 3.00 (0.019)
  Overall Plaque Score after 6 weeks | 2.65 (0.030) | 2.98 (0.021)
  Overall Plaque Score after 12 weeks | 2.55 (0.029) | 2.92 (0.025)
  Overall Plaque Score after 24 weeks | 2.52 (0.032) | 2.95 (0.020)
  Interproximal Plaque Score at Baseline | 3.12 (0.019) | 3.08 (0.018)
  Interproximal Plaque Score after 6 weeks | 2.73 (0.029) | 3.05 (0.020)
  Interproximal Plaque Score after 12 weeks | 2.64 (0.028) | 3.01 (0.022)
  Interproximal Plaque Score after 24 weeks | 2.61 (0.031) | 3.03 (0.019)

ADVERSE EVENTS:
Arm/Group | Sodium Bicarbonate Dentrifice | 0% Sodium Bicarbonate Dentrifice
Serious Adverse Events (participants affected / at risk) | 0/124 | 0/123
Other Adverse Events (participants affected / at risk) | 7/124 | 8/123
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sodium Bicarbonate Dentrifice (N=124) | 0% Sodium Bicarbonate Dentrifice (N=123)
MOUTH INJURY (Injury, poisoning and procedural complications) | 3 | 3
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 1 | 1
THERMAL BURN (Injury, poisoning and procedural complications) | 1 | 1
BRONCHITIS (Infections and infestations) | 1 | 0
NASOPHARYNGITIS (Infections and infestations) | 0 | 1
OVARIAN CYST RUPTURED (Respiratory, thoracic and mediastinal disorders) | 1 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 1
GINGIVAL PAIN (Gastrointestinal disorders) | 0 | 1
SENSITIVITY OF TEETH (Gastrointestinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.